CLINICAL TRIAL: NCT06570421
Title: 24-months, Open-label, Single-Site Extension Study to Evaluate Safety, Tolerability and Efficacy of the Home-based Peroneal Electrical Transcutaneous NeuroModulation (Peroneal eTNM®) Treatment Via Nerve Stimulator URIS ITM in Treatment of Symptoms Related to Movement Disorders in Subjects With Parkinson's Disease (PD) and Essential Tremor (ET)
Brief Title: 24-months Study to Evaluate Safety and Efficacy of Peroneal Transcutaneous NeuroModulation in Subjects With Parkinson's Disease and Essential Tremor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stimvia s.r.o. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS005
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease; Essential Tremor
Keywords: Parkinson Diseases (PD); Essential Tremor (ET); Peroneal Electrical Transcutaneous Neuromodulation; pETNM
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peroneal eTNM arm (Experimental): All patients will receive treatment with peroneal eTNM
  Interventions: Device: Peroneal electrical transcutaneous neuromodulation (peroneal eTNM®)

INTERVENTIONS:
Device: Peroneal electrical transcutaneous neuromodulation (peroneal eTNM®) — This is a non-invasive intervention, which utilizes direct transcutaneous, electrical stimulation of the peroneal nerve
  Other Names: URIS

SUMMARY:
This study investigates the long-term safety and tolerability of home peroneal eTNM® therapy using the URIS I™ device in subjects with Parkinson's disease (PD) or Essential Tremor (ET). Previously, a 6-week open-label pilot study with 24 PD or ET patients demonstrated that home-based peroneal eTNM® is safe, well-tolerated, and has a high adherence rate of over 90%. No treatment-related adverse events were observed. Although the pilot study was not designed to prove efficacy, it suggested positive effects on tremor, with improvements sustained for weeks after treatment. This extension study aims to further evaluate the long-term safety, tolerability, and efficacy of peroneal eTNM® in PD and ET patients.

DETAILED DESCRIPTION:
This is a study to investigate the long-term safety and tolerability of home peroneal eTNM® delivered by URIS I™ in subjects with PD or ET. The safety, tolerability and efficacy of the home-based peroneal eTNM® using URIS ITM neurostimulator in the treatment of symptoms related to movement disorders in subjects with PD and ET has been recently investigated in the study (NTC06036368). This 6-weeks, open-label, single-site pilot study enrolled 24 patients with either PD or ET and was completed in April 2024. This pilot study showed that home-based peroneal eTNM® was safe and well tolerated by patients. No adverse events related to treatment were observed during the study period. These data confirm the excellent safety profile of the peroneal eTNM® that has been observed in previous studies in the overactive bladder population. In addition, all patients were able to stimulate themselves at home without assistance. Adherence to the treatment was very high, reaching well over 90 %. Although this pilot study was not designed to demonstrate the efficacy of peroneal eTNM®, due to its pilot nature and the small sample size, the observed results suggest noteworthy positive effects on rest, postural and kinetic tremor as measured visually, by accelerometers and by validated MDS-UPDRS and TETRAS scales. Importantly, patients reported sustained improvement in tremor throughout the treatment and continuously for several weeks after conclusion of the 6 weeks stimulation period. Data obtained at EoS visit (6 weeks after the last stimulation) lend support for a long-lasting persistence of the effect. Based on these data, the present extension study is designed to evaluate the long-term safety, tolerability and efficacy of peroneal eTNM® in patients with PD and ET. The study will use the medical device URIS I™, which has been assessed for conformity and issued a declaration of conformity. This agent will be used for a different indication, or on a different group of patients, however, without any change in the procedure of use. The clinical trial will be conducted in accordance with clinical trial plan TS005.

ELIGIBILITY:
Inclusion Criteria:

* Has completed participation in study TS004-PD
* Competent and willing to provide written, informed consent to participate in the study.
* Stable dose of any chronic medications, if applicable, for 30 days prior to study entry
* Willing to comply with study protocol requirements.
* Subject agrees not to participate in another study from 30 days prior the baseline visit until the final study visit.
* For subjects with PD:

  * Bradykinesia in "on" period based on clinical assessment
  * Rigidity in "on" period based on clinical assessment
  * Hand/arm exhibiting tremor (resting and/or intentional and/or postural) ≥ grade 1 as assessed by the MDS-UPDRS tremor score in "on" period
* For subjects with ET:

  * Visible hand/arm and/or foot/leg tremor (resting and/or intentional and/or postural) ≥ grade 1 as assessed by the TETRAS

Exclusion Criteria:

* Implanted electrical medical device, such as a pacemaker, defibrillator, or deep brain stimulator
* Suspected or diagnosed epilepsy or other seizure disorder
* Presence of clinical signs or diagnosis of dementia
* Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at stimulation site
* Presence of clinical signs of peripheral neuropathy on lower limbs
* Presence of chorea and/or dyskinesia
* Clinical symptoms or diagnosis of major depressive disorder
* Presence of any other neurodegenerative disease. These may include multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease.
* Botulinum toxin injection within 6 months prior to study enrollment
* Subject is breastfeeding, pregnant, intends to become pregnant during the study, or of childbearing potential, sexually active and not practicing a highly reliable method of birth control (these are methods with a failure quotient of <1% year such as hormonal implants, injectable contraceptives, oral contraceptives of combination type, intra-uterine pessaries restricted to hormone contraceptive coil, sexual abstinence or vasectomy of the partner). The pregnancy test in urine at Visits 1 needs to be negative in women of childbearing potential.
* Subjects unable to communicate effectively with the investigator and staff
* Life expectancy less than 6 months
* Subject with active malignant disease
* Subject who, in the opinion of the physician, may interfere with optimal participation in the clinical trial or may pose a risk to the subject
* Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability Assessed by Treatment Emergent Adverse Events | Baseline to end of the treatment (24 months, based on the study protocol)
  Safety and tolerability based on all safety data collected in the study, including number and type of treatment emergent adverse events (TRAEs).

SECONDARY OUTCOMES:
Therapy Response Measured by Patient Global Impression of Improvement (PGI-I) Scale | Baseline to end of the treatment (24 months, based on the study protocol)
  Change in Patient Global Impression of Improvement scale (Scores 1-7, lower number = better)

OTHER OUTCOMES:
Exploratory endpoints | Baseline to end of the treatment (24 months, based on the study protocol)
  The Movement Disorders Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) score (both total score and subscores) (applicable only for subjects with PD)(0-260, lower score = better)
Exploratory endpoints | Baseline to end of the treatment (24 months, based on the study protocol)
  Essential tremor rating assessment scale (TETRAS) score (applicable only for subjects with ET, 0-64, lower scores = better))
Exploratory endpoints | Baseline to end of the treatment (24 months, based on the study protocol)
  Tremor intensity measured visually (including camera recordings) in millimetres (a higher number = a more intensive tremor)
Exploratory endpoints | Baseline to end of the treatment (24 months, based on the study protocol)
  Quality of life measured by European Quality of Life-5 Dimensions questionnaire (EQ-5D-5L)(0.532-1.000, higher score = better)
Exploratory endpoints | Baseline to end of the treatment (24 months, based on the study protocol)
  Quality of Life in Essential Tremor Questionnaire (QUEST) - applicable only for subjects with ET (0 - 100, lower score better)
Exploratory endpoints | Baseline to end of the treatment (24 months, based on the study protocol)
  Safety assessments:
  * Adverse events (AEs)
  * Treatment-emergent adverse events (TRAEs)
  * Serious adverse events (SAEs)
  * Serious adverse device effects (SADEs) - both anticipated SADEs (ASADEs) and unanticipated SADEs (USADEs)
Exploratory endpoints | Baseline to end of the treatment (24 months, based on the study protocol)
  Patient satisfaction using the Treatment Satisfaction Visual Analog scale (TS-VAS)(0-100, higher score = better)
Exploratory endpoints | Baseline to end of the treatment (24 months, based on the study protocol)
  Disease-specific quality of life measured by Parkinson's Disease Questionnaire (PDQ -39)(0-100, lower score = better)

CONTACTS AND LOCATIONS:
Overall Officials: David Skoloudik, MD, Ph.D., Principal Investigator — Cerebrovaskularni poradna s.r.o.
Locations (1):
- Cerebrovaskulární poradna s.r.o., Ostrava, Czechia

IPD SHARING:
Plan to Share IPD: No